CLINICAL TRIAL: NCT06705985
Title: Treatment of Lateral Knee Joint Pain with Artificial Lateral Meniscus Prosthesis After Meniscectomy
Brief Title: Early Artificial Lateral Prosthesis
Acronym: EARTH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ATRO Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AM-101
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Post-Meniscectomy Pain Syndrome
Keywords: meniscus; lateral; prosthesis

STUDY DESIGN:
Intervention Model Description: The objective of the clinical investigation is to evaluate the safety and performance of the LMP system and to demonstrate that the system is able to replace the function of the natural meniscus to provide pain relief in the lateral compartment of the meniscus-deficient knee. No formal hypothesis testing will be conducted, given the feasibility design of this clinical investigation.
  Evaluation of safety of the LMP system will occur throughout the investigation with the reporting of the nature and frequency of all adverse events observed during the clinical investigation and their timing, severity and relatedness to the investigational device or procedure. In addition, the incidence and nature of secondary surgical intervention will be assessed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lateral Meniscus Prosthesis (Experimental): Implantation of the Lateral Meniscus Prosthesis, intended to replace the function of the natural meniscus to provide unicompartmental pain relief in the meniscus-deficient knee.
  Interventions: Device: Implantation of lateral meniscus prosthesis

INTERVENTIONS:
Device: Implantation of lateral meniscus prosthesis — Implantation of a lateral meniscus prosthesis after meniscectomy.

SUMMARY:
The device subject to this clinical investigation has been developed for treating patients with a history of partial or total meniscectomy, who suffer from symptomatic unicompartmental pain in the meniscus-deficient knee: the post-meniscectomy pain syndrome. The intended purpose of the system is to replace the lateral native meniscus and its function after meniscectomy by distributing tibio-femoral loads and provide a clinically relevant reduction of pain and improvement of joint function.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 18 to 70 years (inclusive) at the time of screening
2. Has a history of partial or total meniscectomy
3. Has post-meniscectomy pain syndrome (defined as symptomatic unicompartmental pain in the meniscus- deficient knee without severe cartilage damage- Kellgren & Lawrence grade 3-4) in the lateral compartment as confirmed by patient history and MRI
4. Has a KOOS Pain of ≤ 75 at the time of screening
5. Failed conservative treatment options (non-operative treatments of the knee, i.e., self-management exercise programs, physical therapy, braces, pain medication, and intra-articular corticosteroids)
6. Has neutral alignment < ± 3° of the mechanical axis
7. Is willing to be implanted with the LMP System and to comply with instruction for use
8. Is able and willing to do the study required follow-up visits, questionnaires, X-rays, and MRI
9. Is able and willing to understand and sign the study Informed Consent Form
10. Is able to read and understand the national language of the country in which the clinical site is located

Exclusion Criteria:

1. Has progressed knee osteoarthritis, Kellgren & Lawrence grade 3- 4 in the lateral compartment
2. Has evidence of a modified Outerbridge Grade IV cartilage loss on the lateral tibial plateau or femoral condyle that potentially could contact the meniscus prosthesis
3. Has medial compartment pain and Grade III or Grade IV modified Outerbridge cartilage score in the medial compartment
4. Has a varus or valgus knee deformity of > 3°
5. Has a valgus alignment that is not passively correctable
6. Has a laxity level of more than Grade II (IKDC), primary or secondary to an injury of the anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or lateral collateral ligament (LCL) and/or medial collateral ligament (MCL)
7. Has significant trochlear dysplasia, patellar instability or symptomatic patellar misalignment
8. Has patellar compartment pain and Grade III or Grade IV modified Outerbridge cartilage score in the patellar compartment
9. Had an ACL reconstruction performed < 9 months prior to surgery
10. Has a BMI > 35 at the time of screening
11. Received any type of prosthetic knee implant made of artificial non-resorbable plastic, metal or ceramic, not including the lateral meniscus prosthesis
12. Has a knee flexion contracture > 10°
13. Has flexion < 90°
14. Had a knee alignment correction osteotomy < 9 months ago
15. Has insufficiency fractures or avascular necrosis of the lateral compartment
16. Has an active infection or tumor (local or systemic)
17. Has any type of knee joint inflammatory disease including Sjogren's syndrome
18. Has neuropathic knee osteoarthropathy, also known as Charcot joint
19. Has any medical condition that does not allow possible arthroscopy of the knee
20. Has neurological deficit (sensory, motor, or reflex)
21. Anticipates having another lower extremity surgery during the study period
22. Is contraindicated for corticosteroid injections (i.e., patients with allergy to any of the components or with idiopathic thrombocytopenic purpura)
23. Has received any corticosteroid knee injections ≤ 3 months prior to surgery
24. Has proven osteoporosis
25. Is on immunostimulating or immunosuppressing agents
26. Has ipsilateral or contralateral lower limb joint conditions that may affect ambulation or study outcomes (e.g. have a leg length discrepancy > 2.5 cm [1 inch], causing a noticeable limp)
27. Is a female who is lactating, expecting, or is intending to become pregnant during the study period
28. Is an active smoker at the time of surgery
29. Is mentally incapacitated (incapable of appraising or controlling conduct) or have mental disability (e.g., dementia or Alzheimer's)
30. Has a condition or be in a situation that, in the Investigator's opinion, may confound the clinical investigation results, may risk the safety of the patient, or may interfere significantly with the subject's participation in the clinical investigation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-21 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 12 months after implantation.
  Adverse events within 12 months after implantation.
Implant integrity | 12 months after implantation.
  Assessed by MRI.

SECONDARY OUTCOMES:
KOOS | 24 months.
  KOOS (overall including all subscales) at 6 weeks, 3, 6, 12, 24 months.
Lysholm | 24 months.
  Lysholm scale at 6 weeks, 3, 6, 12, 24 months.
OKS | 24 months.
  OKS at 6, 12, 24 months.
EQ-5D-5L | 24 months.
  EQ-5D-5L at 6, 12, 24 months.
WORQ | 24 months.
  WORQ at 6 weeks, 3, 6, 12, 24 months.
SF-36 | 24 months.
  SF-36 at 6, 12, 24 months.
Likert - Patient satisfaction | 24 months.
  Patient satisfaction on a 5-point Likert scale at 6, 12, 24 months.
Tegner Activity Scale | 24 months.
  Tegner Activity Scale at 6 weeks, 3, 6, 12, 24 months.
IKDC Knee Examination Form | 24 months.
  IKDC Knee Examination Form at screening, surgery, 6 weeks, 3, 6, 12, 24 months.
Knee X-ray (weight-bearing) | 24 months.
  Knee X-ray (weight-bearing) at 6, 12, and 24 months to evaluate the height of the joint space.
Knee X-ray (weight-bearing, long-leg) | 24 months.
  • Knee X-ray (weight-bearing, long-leg) at 6, 12, and 24 months to evaluate the mechanical axis.
Knee X-ray (non-weight-bearing, supine) | 24 months.
  Knee X-ray (non-weight-bearing, supine) at 12, and 24 months to evaluate the mechanical axis.
Knee MRI (non-weight-bearing) | 24 months.
  Knee MRI (non-weight-bearing) at implantation surgery (+(within
  1 week, preferably peroperative), 6, 12, and 24 months for implant and joint integrity (cartilage status) assessment (including focal defects, bone marrow lesions, and bone tunnels/fixation sites).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands